CLINICAL TRIAL: NCT01993134
Title: Efficacy Assessment of Two Antibiotic Prophylaxis Regimens in Oral and Maxillofacial Trauma Surgery.
Acronym: EAPRTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Giordano Bruno Paiva Campos, DDS, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ATB-001
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Facial Fractures
Keywords: Postoperative infection; Antibiotic prophylaxis; Cefazolin
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefazolin (Experimental): 2g of Cefazolin, 20minutes before sugery. After surgery, 1g of cefazolin 06/06h.
  Interventions: Procedure: Cefazolin
- Cefazolin Single Dose (Active Comparator): 2g of Cefazolin, 20minutes before sugery. After surgery, no drugs.
  Interventions: Procedure: Cefazolin Single Dose

INTERVENTIONS:
Procedure: Cefazolin — Cefazolin, 2g/IV, prior to surgery, and after surgery recieved 4 aditional doses 1g/IV of Cefazolin.
  Arms: Cefazolin
Procedure: Cefazolin Single Dose — Patients received 2g of Cefazolin (Cefazolin Sodium - Ampoule- 1g - Genéricos Brasil), administered intravenously but none was administered in the post-operative period
  Arms: Cefazolin Single Dose

SUMMARY:
The study set out to evaluate the efficacy of two antibiotic prophylaxis regimens in patients with facial fractures admitted to the Oral and Maxillofacial Surgery and Traumatology services of the Onofre Lopes University Hospital attached to the Federal University of Rio Grande do Norte.

DETAILED DESCRIPTION:
The study set out to evaluate the efficacy of two antibiotic prophylaxis regimens in patients with facial fractures admitted to the Oral and Maxillofacial Surgery and Traumatology services of the Onofre Lopes University Hospital attached to the Federal University of Rio Grande do Norte.This clinical study was prospective, randomized and controlled. Patients underwent surgery for facial fracture reduction and fixation under general anesthetic. Prior to surgery, patients were randomly divided into two groups. Group 1 patients each received 2g of Cefazolin (Cefazolin Sodium - Ampoule- 1g - Genéricos Brasil), administered intravenously but none was administered in the post-operative period. Group II patients received the same dose prior to the operation but in the post-operative period they also received 4 additional 1 g doses of Cefazolin intravenously, completing a 24 period of antibiotic prophylaxis. In the case of operations that lasted for more than 4 hours, an additional 1g dose was given.

The surgical operations involved intra and extra-oral interventions and when required internal rigid fixation was undertaken using titanium plates and screws. Patients were given advice on oral hygiene procedures to be followed in the post-operative period that included chlorhexidine (0.12%) oral rinses and care to be taken with the surgical wounds.

Post-operative follow up was conducted in the 1st, 2nd, 4th and 6th weeks. The criteria used to determine the presence of infection were: a) pus drainage at the fracture site or in the vicinity of the surgical intervention site; b) increased swelling 7 days after the operation; c) presence of a fistula in the area of the surgical intervention or at the site of the fracture, with active drainage; d) other clinical features observed by the evaluator including typical signs of infection such as fever, edema, and localized redness.

Descriptive analysis was made of the independent variables, namely, age, sex, presence of systemic diseases, trauma cause, drug use (tobacco, alcohol, marijuana, crack, cocaine , etc.), the time lapse between the trauma event and the surgical operation, length of the operation, and the measures adopted when infections were detected.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* ASA I, II, III
* have facial fractures, that request surgical treatement, and whitout infection

Exclusion Criteria:

* Patients with pan-facial fractures
* Or requiring surgery longer than six hours

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of postoperative infection | 45 days
  Post-operative follow up was conducted in the 1st, 2nd, 4th and 6th weeks. The criteria used to determine the presence of infection were: a) pus drainage at the fracture site or in the vicinity of the surgical intervention site; b) increased swelling 7 days after the operation; c) presence of a fistula in the area of the surgical intervention or at the site of the fracture, with active drainage; d) other clinical features observed by the evaluator including typical signs of infection such as fever, edema, and localized redness.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Germano, PhD, Study Chair — Universidade Federal do Rio Grande do Norte
Locations (1):
- Oral and Maxillofacial Surgery and Traumatology services of the Onofre Lopes University Hospital, Natal, Rio Grande do Norte, Brazil